CLINICAL TRIAL: NCT01623869
Title: Phase II Study of the Angiopoietin-1 and -2 Peptibody AMG 386 for the Treatment of Angiosarcoma
Brief Title: Trebananib in Treating Patients With Advanced Angiosarcoma That Cannot Be Removed by Surgery
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NCI-2012-01978; NCI-2012-01978 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); CDR0000735380; CALGB-A091103; A091103 (Other: Alliance for Clinical Trials in Oncology); A091103 (Other: CTEP); U10CA180821 (NIH); U10CA031946 (NIH)
Record Dates: First submitted 2012-06-17; First posted 2012-06-20 (Estimated); Results first posted 2015-07-02 (Estimated); Last update posted 2015-10-19 (Estimated); Status verified 2015-06

CONDITIONS: Adult Angiosarcoma; Recurrent Adult Soft Tissue Sarcoma; Stage III Adult Soft Tissue Sarcoma; Stage IV Adult Soft Tissue Sarcoma
MeSH Terms: conditions — Hemangiosarcoma; Sarcoma | interventions — trebananib

ARMS (1):
- Treatment (trebananib) (Experimental): Patients receive 30 mg/kg trebananib IV over 30-60 minutes on days 1, 8, 15, and 22. Courses repeat every 28 days in the absence of disease progression or unacceptable toxicity.
  Interventions: Other: Laboratory Biomarker Analysis; Biological: Trebananib

INTERVENTIONS:
Other: Laboratory Biomarker Analysis — Correlative studies
Biological: Trebananib — Given IV
  Other Names: AMG 386; Angiopoietin 1/2-Neutralizing Peptibody AMG 386

SUMMARY:
This phase II trial studies how well trebananib works in treating patients with advanced angiosarcoma that cannot be removed by surgery. Trebananib may stop the growth of tumor cells by blocking blood flow to the tumor.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To determine the overall response rate (ORR), defined as complete response (CR) +partial response (PR), in patients with advanced, unresectable angiosarcoma treated with trebananib (AMG 386).

SECONDARY OBJECTIVES:

I. To evaluate the progression-free survival (PFS) and overall survival (OS) of patients with advanced, unresectable angiosarcoma treated with AMG 386.

TERTIARY OBJECTIVES:

I. To correlate ORR, PFS, and OS with: Baseline and post-treatment changes in expression of angiopoietin 2 (Ang2) and TEK tyrosine kinase, endothelial (Tie2) by immunohistochemistry (IHC); Serum levels of angiopoietin 1 (Ang1) and Ang2; Baseline and post-treatment changes in phospho-receptor tyrosine kinase status of TIE2, vascular endothelial growth factor receptor 2 (VEGFR-2), phosphatidylinositol 3 kinase (PI3K), mitogen-activated protein kinase Inhibitor (MEK) in tumor tissue; Mutational status of VEGFR-2 and amplification of v-myc myelocytomatosis viral oncogene homolog (avian) (MYC)/fms-related tyrosine kinase 4 (FLT4).

OUTLINE:

Patients receive trebananib intravenously (IV) over 30-60 minutes on days 1, 8, 15, and 22. Courses repeat every 28 days in the absence of disease progression or unacceptable toxicity.

After completion of study treatment, patients are followed up for 4 weeks and then every 6 months for 18 months.

ELIGIBILITY:
Inclusion Criteria:

* Patients must have histologically confirmed angiosarcoma that is unresectable
* Patients must have measurable disease per Response Evaluation Criteria in Solid Tumors(RECIST) 1.1, defined as at least one lesion that can be accurately measured in at least one dimension (longest diameter to be recorded for non-nodal lesions and short axis for nodal lesions) as >= 2 cm with conventional techniques or as >= 1 cm with spiral computed tomography (CT) scan, magnetic resonance imaging (MRI), or calipers by clinical exam
* Patients must have had =< 4 prior systemic treatment regimens
* Eastern Cooperative Oncology Group (ECOG) 0-1 or Karnofsky >= 70%
* Life expectancy of greater than 3 months
* Leukocytes >= 3,000/mcL
* Absolute neutrophil count >= 1,500/mcL
* Hemoglobin >= 8.5g/dL
* Platelet count >= 60,000/mcL
* Total bilirubin =< 1.5 times institutional upper limit of normal (ULN)
* Aspartate aminotransferase (AST)(serum glutamic oxaloacetic transaminase [SGOT]) =< 2.5 times institutional ULN
* Alanine aminotransferase (ALT) (serum glutamic pyruvate transaminase[SGPT]) =< 2.5 times institutional ULN
* Partial thromboplastin time (PTT) or activated (a)PTT =< 1.5 times ULN per institutional laboratory range
* International normalized ratio(INR) =< 1.5 (unless on warfarin)
* Creatinine =< 1.5 times ULN OR creatinine clearance > 40 mL/min per 24-hour urine collection or calculated according to the Cockcroft-Gault formula
* Urinary protein =< 30 mg/dL in urinalysis or =< 1+ on dipstick, unless quantitative protein is < 1,000 mg in a 24-hour urine sample
* Women of childbearing potential and men must agree to use adequate contraception (hormonal or barrier method of birth control; abstinence) prior to study entry and for the duration of study participation

  * Women of child-bearing potential and men must agree to use adequate contraception (hormonal or barrier method of birth control; abstinence) prior to study entry and for the duration of study participation should a woman become pregnant or suspect she is pregnant while she or her partner is participating in this study, she should inform her treating physician immediately
  * Breastfeeding must be discontinued if the mother is treated with AMG 386; these potential risks may also apply to other agents used in this study
  * Female of childbearing potential is defined as the following: A female of childbearing potential is a sexually mature woman who: 1) has not undergone a hysterectomy or bilateral oophorectomy or 2) has not been naturally postmenopausal (amenorrhea following cancer therapy does not rule out childbearing potential) for at least 24 consecutive months (i.e., has had menses at any time in the preceding 24 consecutive months)
* Generally well-controlled blood pressure with systolic blood pressure =< 150 mm Hg and diastolic blood pressure =< 90 mm Hg (Note: The use of anti-hypertensive medications to control hypertension is permitted)
* Ability to understand and the willingness to sign a written informed consent document

Exclusion Criteria:

* No known history of brain metastases
* History of clinically significant bleeding within 6 months of enrollment/randomization
* No unresolved toxicities from prior systemic therapy that are Common Terminology Criteria for Adverse Events (CTCAE) version 4.0 >= grade 2 in severity except alopecia
* Currently or previously treated with AMG 386, or other molecules that inhibit the angiopoietins or Tie2 receptor
* Clinically significant cardiovascular disease within 12 months prior to enrollment/randomization, including myocardial infarction, unstable angina, grade 2 or greater (CTCAE version 4.0) peripheral vascular disease, cerebrovascular accident, transient ischemic attack, congestive heart failure, or arrhythmias not controlled by outpatient medication or placement of percutaneous transluminal coronary angioplasty/stent
* Major surgery within 28 days prior to enrollment or still recovering from prior surgery
* Treatment within 30 days prior to enrollment with strong immune modulators including, but not limited to, systemic cyclosporine, tacrolimus, sirolimus, mycophenolate mofetil, methotrexate, azathioprine, rapamycin, thalidomide, lenalidomide, and targeted immune modulators such as abatacept (CTLA-4- -Ig),adalimumab, alefacept, anakinra, belatacept (LEA29Y), efalizumab, etanercept, infliximab, or rituximab
* Non-healing wound
* Subject not consenting to the use of highly effective contraceptive precautions (e.g., double barrier method [i.e., condom plus diaphragm]) during the course of the study and for 6 months after administration of the last study medication
* History of allergic reactions attributed to compounds of similar chemical or biologic composition to AMG 386
* History of allergic reactions to bacterially-produced proteins
* Patients who have had chemotherapy or radiotherapy within 4 weeks (6 weeks for nitrosoureas or mitomycin C) prior to entering the study or those who have not recovered from adverse events due to agents administered more than 4 weeks earlier
* Patients who have not yet completed at least 21 days (30 days for prior monoclonal antibody therapy) since ending other investigational device or drug trials, or who are currently receiving other investigational treatments
* Uncontrolled intercurrent illness including, but not limited to, ongoing or active infection, symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia, or psychiatric illness/social situations that would limit compliance with study requirements
* Non-pregnant, non-nursing; Note: Women of child bearing potential must have a pregnancy test, serum based within 7 days prior to registration; this is because AMG 386 is an inhibitor of angiogenesis with the potential for teratogenic or abortifacient effects
* Patients with a history of venous or arterial thromboembolism within 12 months prior to enrollment/randomization should be excluded

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 16 (Actual)
Dates: Start 2012-07; Primary Completion 2014-09 (Actual); Study Completion 2015-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Sandra D'Angelo, Principal Investigator — Alliance for Clinical Trials in Oncology
Locations (70):
- United States (70):
  - Beebe Medical Center, Lewes, Delaware
  - Christiana Care Health System-Christiana Hospital, Newark, Delaware
  - Washington Hospital Center, Washington D.C., District of Columbia
  - Oncare Hawaii Inc-POB II, Honolulu, Hawaii
  - Queen's Medical Center, Honolulu, Hawaii
  - Straub Clinic and Hospital, Honolulu, Hawaii
  - University of Hawaii Cancer Center, Honolulu, Hawaii
  - Oncare Hawaii Inc-Kuakini, Honolulu, Hawaii
  - Kapiolani Medical Center for Women and Children, Honolulu, Hawaii
  - Castle Medical Center, Kailua, Hawaii
  - Wilcox Memorial Hospital and Kauai Medical Clinic, Lihue, Hawaii
  - Oncare Hawaii Inc-Pali Momi, ‘Aiea, Hawaii
  - Pali Momi Medical Center, ‘Aiea, Hawaii
  - Saint Joseph Medical Center, Bloomington, Illinois
  - Illinois CancerCare-Bloomington, Bloomington, Illinois
  - Graham Hospital Association, Canton, Illinois
  - Illinois CancerCare-Canton, Canton, Illinois
  - Illinois CancerCare-Carthage, Carthage, Illinois
  - Memorial Hospital, Carthage, Illinois
  - Northwestern University, Chicago, Illinois
  - Eureka Hospital, Eureka, Illinois
  - Illinois CancerCare-Eureka, Eureka, Illinois
  - Illinois CancerCare Galesburg, Galesburg, Illinois
  - Illinois CancerCare-Havana, Havana, Illinois
  - Mason District Hospital, Havana, Illinois
  - Illinois CancerCare-Kewanee Clinic, Kewanee, Illinois
  - Illinois CancerCare-Macomb, Macomb, Illinois
  - Mcdonough District Hospital, Macomb, Illinois
  - Holy Family Medical Center, Monmouth, Illinois
  - Illinois CancerCare-Monmouth, Monmouth, Illinois
  - Bromenn Regional Medical Center, Normal, Illinois
  - Community Cancer Center Foundation, Normal, Illinois
  - Illinois CancerCare-Community Cancer Center, Normal, Illinois
  - Illinois CancerCare-Ottawa Clinic, Ottawa, Illinois
  - Ottawa Regional Hospital and Healthcare Center, Ottawa, Illinois
  - Illinois CancerCare-Pekin, Pekin, Illinois
  - Pekin Cancer Treatment Center, Pekin, Illinois
  - Methodist Medical Center of Illinois, Peoria, Illinois
  - Proctor Hospital, Peoria, Illinois
  - Illinois CancerCare-Peoria, Peoria, Illinois
  - Illinois Oncology Research Association CCOP, Peoria, Illinois
  - OSF Saint Francis Medical Center, Peoria, Illinois
  - Illinois CancerCare-Peru, Peru, Illinois
  - Illinois Valley Hospital, Peru, Illinois
  - Illinois CancerCare-Princeton, Princeton, Illinois
  - Perry Memorial Hospital, Princeton, Illinois
  - Illinois CancerCare-Spring Valley, Spring Valley, Illinois
  - Carle Cancer Center, Urbana, Illinois
  - Franciscan Saint Francis Health-Indianapolis, Indianapolis, Indiana
  - Reid Hospital and Health Care Services, Richmond, Indiana
  - University of Iowa/Holden Comprehensive Cancer Center, Iowa City, Iowa
  - Siouxland Regional Cancer Center, Sioux City, Iowa
  - Mercy Medical Center-Sioux City, Sioux City, Iowa
  - Saint Luke's Regional Medical Center, Sioux City, Iowa
  - Union Hospital of Cecil County, Elkton MD, Maryland
  - Mayo Clinic, Rochester, Minnesota
  - Washington University School of Medicine, St Louis, Missouri
  - Cooper Hospital University Medical Center, Camden, New Jersey
  - Memorial Sloan-Kettering Cancer Center, New York, New York
  - Grandview Hospital, Dayton, Ohio
  - Good Samaritan Hospital - Dayton, Dayton, Ohio
  - Miami Valley Hospital, Dayton, Ohio
  - Samaritan North Health Center, Dayton, Ohio
  - Dayton CCOP, Dayton, Ohio
  - Blanchard Valley Hospital, Findlay, Ohio
  - Atrium Medical Center-Middletown Regional Hospital, Franklin, Ohio
  - Wayne Hospital, Greenville, Ohio
  - Kettering Medical Center, Kettering, Ohio
  - Upper Valley Medical Center, Troy, Ohio
  - Greene Memorial Hospital, Xenia, Ohio

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Treatment (Trebananib)
Started | 16
Completed | 16
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Treatment (Trebananib)
Number analyzed (Participants) | 16
Age, Continuous [Median (Full Range); unit: years] | 68.5 [24 to 91]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 10
  Male | 6
Region of Enrollment [Number; unit: participants]
  United States | 16

OUTCOME MEASURES:

1. Primary Outcome: Confirmed Response Rate (CR or PR) Using RECIST
Description: Response and progression will be evaluated using the international RECIST guidelines (v1.1). Patients are evaluated every 8 weeks for disease status, with a subsequent 4 week assessment required to confirm a response.
  Complete Response (CR) - All of the following must be true:
  1. Disappearance of all target and non-target lesions,
  2. Each target lesion and non-target lymph node must have reduction in short axis to <1.0 cm.
  Partial Response (PR):
  1. At least a 30% decrease from the baseline measurements of the sum of the longest diameter for all target lesions plus the sum of the short axis of all the target lymph nodes at current evaluation.
  2. Persistence of one or more non-target lesions or non-target lymph nodes. The confirmed response rate is estimated as the number of patients having a CR or PR, divided by the number of eligible patients having at least one post-baseline assessment. The 95% confidence intervals provided using the method of Duffy and Santner.
Time Frame: Up to 18 months
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Treatment (Trebananib)
Number analyzed (Participants) | 16
percentage of participants | 0 [0 to 20.6]

2. Secondary Outcome: Progression Free Survival (PFS)
Description: Progression-free survival (PFS) is defined as the duration of time from the start of treatment to time of radiologic or clinical progression or death, whichever occurs first. PFS will be censored at most recent radiographic assessment date for patients remaining alive at the time of the statistical analysis. Kaplan-Meier methodology will be used to estimate the distribution of PFS.
Time Frame: From the start of treatment to time of radiologic or clinical progression or death, whichever occurs first, assessed up to 18 months
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Treatment (Trebananib)
Number analyzed (Participants) | 16
months | 1.6 [1.4 to 1.7]

3. Secondary Outcome: OS
Description: Overall survival (OS) is the duration of time from the date of registration/randomization to the date of death or the date of last follow-up for patients who remain alive or who are lost to follow-up at the time of the analysis. Kaplan-Meier methodology will be used to estimate the distribution of OS.
Time Frame: From the date of registration to the date of death or the date of last follow-up, assessed up to 18 months
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Treatment (Trebananib)
Number analyzed (Participants) | 16
months | 6.4 [4.0 to 11.1]

ADVERSE EVENTS:
Time Frame: Evaluated monthly from the date of randomization until 30 days following a patient's last dose.
Description: Maximum severity per AE classification is reported, per patient.
Arm/Group | Treatment (Trebananib)
Serious Adverse Events (participants affected / at risk) | 6/16
Other Adverse Events (participants affected / at risk) | 12/16
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Treatment (Trebananib) (N=16)
Cardiac arrest (Cardiac disorders) | 1 (1)
Wound infection (Infections and infestations) | 1 (1)
Activated partial thromboplastin time prolonged (Investigations) | 1 (1)
Hypocalcemia (Metabolism and nutrition disorders) | 1 (1)
Hyponatremia (Metabolism and nutrition disorders) | 1 (1)
Chest wall pain (Musculoskeletal and connective tissue disorders) | 1 (1)
Syncope (Nervous system disorders) | 1 (1)
Cough (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Hematoma (Vascular disorders) | 1 (1)
Thromboembolic event (Vascular disorders) | 2 (3)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Treatment (Trebananib) (N=16)
Anemia (Blood and lymphatic system disorders) | 3 (4)
Mucositis oral (Gastrointestinal disorders) | 1 (1)
Nausea (Gastrointestinal disorders) | 2 (2)
Edema face (General disorders) | 2 (6)
Edema limbs (General disorders) | 7 (19)
Fatigue (General disorders) | 3 (3)
Pain (General disorders) | 1 (1)
Allergic reaction (Immune system disorders) | 1 (1)
Infections and infestations - Other, specify (Infections and infestations) | 1 (1)
Urinary tract infection (Infections and infestations) | 1 (1)
Activated partial thromboplastin time prolonged (Investigations) | 2 (6)
Alanine aminotransferase increased (Investigations) | 1 (1)
Alkaline phosphatase increased (Investigations) | 2 (3)
Aspartate aminotransferase increased (Investigations) | 3 (3)
Blood bilirubin increased (Investigations) | 1 (1)
CD4 lymphocytes decreased (Investigations) | 1 (3)
Creatinine increased (Investigations) | 1 (2)
INR increased (Investigations) | 2 (2)
Lymphocyte count decreased (Investigations) | 3 (5)
Platelet count decreased (Investigations) | 2 (4)
Anorexia (Metabolism and nutrition disorders) | 1 (1)
Hyperglycemia (Metabolism and nutrition disorders) | 2 (2)
Hyperkalemia (Metabolism and nutrition disorders) | 1 (1)
Hypoalbuminemia (Metabolism and nutrition disorders) | 3 (7)
Hypocalcemia (Metabolism and nutrition disorders) | 2 (6)
Hypokalemia (Metabolism and nutrition disorders) | 2 (3)
Hyponatremia (Metabolism and nutrition disorders) | 4 (6)
Metabolism and nutrition disorders - Other, specify (Metabolism and nutrition disorders) | 1 (1)
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 (1)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 (1)
Peripheral motor neuropathy (Nervous system disorders) | 1 (2)
Peripheral sensory neuropathy (Nervous system disorders) | 1 (1)
Hematuria (Renal and urinary disorders) | 1 (2)
Cough (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Pulmonary edema (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Periorbital edema (Skin and subcutaneous tissue disorders) | 2 (4)
Rash acneiform (Skin and subcutaneous tissue disorders) | 1 (1)
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 2 (2)
Hypertension (Vascular disorders) | 1 (1)
Lymphedema (Vascular disorders) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less